CLINICAL TRIAL: NCT00056095
Title: Phase II Trial in Intrafamilial Allogeneic Cell Transplant in Patients With Metastatic Kidney Cancer
Brief Title: Allogeneic Stem Cell Transplant in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/0105; FRE-FNCLCC-GETUG-11/0105 (Other: FNCLCC); EU-20234 (Other: European union)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Cyclophosphamide; Cyclosporine; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allograft (compatible family member) (Experimental)
  Interventions: Biological: therapeutic allogeneic lymphocytes; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Procedure: allogeneic bone marrow transplantation; Procedure: peripheral blood stem cell transplantation
- Allograft (compatible non-family member) (Other)
  Interventions: Procedure: allogeneic bone marrow transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes
  Arms: Allograft (compatible family member)
Drug: cyclophosphamide
  Arms: Allograft (compatible family member)
Drug: cyclosporine
  Arms: Allograft (compatible family member)
Drug: fludarabine phosphate
  Arms: Allograft (compatible family member)
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: This phase II trial is studying how well allogeneic stem cell transplant works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 18-month survival rate of patients with metastatic renal cell carcinoma treated with allogeneic stem cell transplantation.
* Determine the objective rate of response of patients treated with this regimen.
* Determine post-transplant immunological reactions and recuperation of patients treated with this regimen.
* Determine the antitumoral activity of this regimen in these patients.

OUTLINE: This is a non-randomized, multicenter study. Patients are assigned to 1 of 2 treatment groups based on availability of a compatible family member for stem cell transplantation.

* Group I: Patients with a compatible family donor receive conditioning chemotherapy comprising cyclophosphamide IV over 2 hours on days -7 and -6 and fludarabine IV once daily on days -5 to -1. Patients undergo filgrastim (G-CSF)-mobilized allogeneic stem cell transplantation on day 0. Patients also receive immunosuppression therapy with cyclosporine beginning on day -2. Patients who have persistent or progressive disease, mixed chimerism, and no evidence of grade 2 or greater graft-vs-host disease, and have been off immunosuppression therapy for 1-2 weeks receive donor lymphocyte infusion on days 7 and 21.
* Group II: Patients without a compatible family donor receive treatment (immunotherapy, vaccination therapy, or chemotherapy) at the discretion of the treating physician.

Patients are followed every 3 months for 5 years.

PROJECTED ACCRUAL: A total of 170 patients (60 patients for group I and 110 patients for group II) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell carcinoma
* No sarcomatoid, pure papillary, or Bellini renal cell cancer
* Measurable and/or evaluable disease
* Disease progression after at least 1 immunotherapy regimen for metastatic disease
* Localized metastases allowed provided the following are true:

  * At least 3 months since prior treatment for metastases
  * Not considered likely to influence outcome of transplantation
* No brain metastases unless treated surgically or radiologically and MRI normal
* Sufficiently healthy, HLA-compatible family member must be available as donor for patients undergoing stem cell transplantation

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Performance status

* ECOG 0-1

Life expectancy

* More than 6 months

Hematopoietic

* Platelet count at least 100,000/mm^3

Hepatic

* Transaminases less than 1.5 times upper limit of normal (ULN)*
* Bilirubin less than 1.5 times ULN* NOTE: *Unless due to Gilbert's disease

Renal

* No renal insufficiency
* Calcium less than 10.4 mg/dL
* Creatinine clearance greater than 50 mL/min

Cardiovascular

* Ejection fraction greater than 50%

Pulmonary

* No DLCO that would preclude fludarabine or busulfan therapy

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No physical obstacle to receiving study treatment
* No known autoimmune disease
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No uncontrolled bacterial, viral, or fungal infection
* No prior or concurrent psychiatric disease
* HIV negative
* HTLV1 negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* No tolerance to fludarabine and busulfan

Endocrine therapy

* No concurrent corticosteroids

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2002-11-04 (Actual); Primary Completion 2008-02-13 (Actual); Study Completion 2016-08-17 (Actual)

PRIMARY OUTCOMES:
Survival rate at 18 months
Objective rate of response
Post-transplant immunological reactions and recuperation
Antitumoral activity

CONTACTS AND LOCATIONS:
Overall Officials: Didier Blaise, MD, Study Chair — Institut Paoli-Calmettes
Locations (26):
- France (26):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - Centre Paul Papin, Angers
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Saint Andre, Bordeaux
  - Chu-Hopital Gabriel Montpied, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU de Grenoble - Hopital Michallon, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Lapeyronie-CHU Montpellier, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital de l'Archet CHU de Nice, Nice
  - Institut Curie Hopital, Paris
  - Hopital Haut Leveque, Pessac
  - Hopital Jean Bernard, Poitiers
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif